CLINICAL TRIAL: NCT00349258
Title: A Prospective Randomized Study Comparing the Use of hCG or GnRH Agonist to Trigger Final Oocyte Maturation in High Responders Undergoing in-Vitro Fertilization Treatment
Brief Title: The Use of GnRH Agonist Trigger in the Prevention of OHSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Organon (Industry)
Organization: UConn Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-277
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2006-07-06 (Estimated); Status verified 2006-02

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: OHSS; PCOS; Previous high response; GnRH antagonist; GnRH agonist; IVF
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Leuprolide

INTERVENTIONS:
Drug: Leuprolide acetate

SUMMARY:
To compare the incidence of ovarian hyperstimulation syndrome (OHSS) and implantation rate between high responder patients using Gonadotropin releasing GnRH) agonist or human chorionic gonadotropin (hCG) to trigger final oocyte maturation.

DETAILED DESCRIPTION:
OHSS is an iatrogenic complication of controlled ovarian hyperstimulation, which in its severe form, may result in significant morbidity. Although, there have been significant advances in in-vitro fertilization (IVF) protocols over the years, the incidence of OHSS have remained stable and there is currently no effective way of preventing this disorder.

hCG is commonly used as a substitute for the endogenous LH surge to induce final oocyte maturation in IVF. Unfortunately, hCG results in a prolonged luteotropic effect because of its long half-life which may result in a potential risk of OHSS in high-risk patients. In contrast, induction of endogenous LH surge with a GnRH agonist may result in a reduced risk of OHSS. This is due both to the shorter half-life of the endogenous LH surge and the subsequent pituitary suppression leading to early luteolysis. However, previous studies have suggested that this approach may impair implantation rates.

There are no randomized studies assessing the effect of GnRH agonist to induce oocyte maturation on the occurrence of OHSS and implantation rates in high-risk patients. The aims of this study are to compare the incidence of OHSS and implantation rates among high-risk patients who used either GnRH agonist or hCG to trigger oocyte maturation after prevention of premature LH surge with either a GnRH antagonist protocol or the dual pituitary suppression protocol, respectively.

High risk patients include women with polycystic ovarian syndrome (PCOS) or PCO morphology (PCOM) on ultrasound without the clinical or biochemical evidence of the syndrome, and patients with previous high response to gonadotropins.

ELIGIBILITY:
Inclusion Criteria:

* age 20-39
* normal early follicular phase serum FSH (≤10.0 IU/l)
* patients with either PCOS or PCOM undergoing their first cycle of IVF or patients with high response in a previous IVF cycle.

Exclusion Criteria:

* Hypogonadotropic hypogonadism

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66
Dates: Start 2004-08; Study Completion 2006-05

PRIMARY OUTCOMES:
OHSS occurrence assessed one week after oocyte retrieval
Implantation rate assessed at seven weeks gestation

SECONDARY OUTCOMES:
Clinical Pregnancy rate assessed at time of ultrasound
Mature oocytes assessed at time of retrieval
Ovarian volume assessed one week after oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Benadiva, MD, Principal Investigator — UConn Health; Lawrence Engmann, MD, Principal Investigator — UConn Health
Locations (1):
- Center for Advanced Reproductive Services, UCHC, Farmington, Connecticut, United States

REFERENCES:
- [Derived] Engmann L, Romak J, Nulsen J, Benadiva C, Peluso J. In vitro viability and secretory capacity of human luteinized granulosa cells after gonadotropin-releasing hormone agonist trigger of oocyte maturation. Fertil Steril. 2011 Jul;96(1):198-202. doi: 10.1016/j.fertnstert.2011.04.071. Epub 2011 May 20. PMID 21601197